CLINICAL TRIAL: NCT00215254
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of Quetiapine in Social Anxiety Disorder
Brief Title: Quetiapine in Social Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5639-04-3R0
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-03

CONDITIONS: Social Anxiety Disorder
Keywords: quetiapine; social anxiety disorder; antipsychotic; pilot study
MeSH Terms: conditions — Phobia, Social | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
The purpose of the study is to examine the effectiveness and tolerability of quetiapine for the treatment of social anxiety disorder (SAD). The hypothesis is that quetiapine will be effective and well-tolerated for patients with social anxiety disorder.

DETAILED DESCRIPTION:
This is an eight week, randomized, double-blind, placebo-controlled trial of quetiapine (100-400 mg/day)in social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients 18-65 years of age
* primary diagnosis of social anxiety disorder, using DSM-IV criteria
* minimum CGI severity score of 4 at baseline
* minimum BSPS score of 20 at baseline
* written informed consent
* negative serum pregnancy test for women of childbearing potential

Exclusion Criteria:

* current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition
* any current primary anxiety disorder other than SAD or current primary depression
* history of substance abuse or dependence with the last 6 months
* suicide risk or serious suicide attempt within the last year
* clinically significant medical condition or laboratory abnormality
* women of childbearing potential who are unwilling to practice an acceptable method of contraception
* concomitant medication use for psychotropic purposes
* history of hypersensitivity to quetiapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-03; Study Completion 2006-02

PRIMARY OUTCOMES:
Brief Social Phobia Scale (BSPS)

SECONDARY OUTCOMES:
Clinical Global Impressions of Severity (CGI-S)
Clinical Global Impressions of Improvement (CGI-I)
Social Phobia Inventory (SPIN)
Hospital Anxiety and Depression Scale (HADS)
Connor Davidson Resilience Scale (CD-RISC)
Sheehan Disability Inventory (SDI)
Barnes Akathisis Scale (BAS)
Simpson-Angus Scale (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States